CLINICAL TRIAL: NCT04923555
Title: Analysis of the Postprandial Effects of a Vegetable Protein Mixture Rich in Arginine, Cysteine and Leucine on Endothelial Dysfunction and Inflammation at Low Noise in Elderly People With Cardiometabolic Risk
Acronym: P-PROBS CM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: RBHP 2021 PICKERING; 2021-A00134-37 (Other: 2021-A00134-37)
Record Dates: First submitted 2021-06-01; First posted 2021-06-11 (Actual); Last update posted 2022-06-13 (Actual); Status verified 2022-06

CONDITIONS: Metabolic Syndrome; Predisposition to Cardiovascular Disease
Keywords: Metabolic syndrome; Endothelial function; Vegetable proteins; Arginine; Cysteine; Leucine; Nutrition assessment; Nutrition physiological phenomena
MeSH Terms: conditions — Metabolic Syndrome | interventions — Plant Proteins, Dietary; Leucine; Arginine; Animal Proteins, Dietary

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Product kit (yogurt) will be labelled and packaged according to the pre-established randomization plane by the pharmacy department of University Hospital of Clermont-Ferrand, France. Kits will be distributed in a blind fashion for each cross over period on the basis of the randomization schedule.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group/Cohort1 (Experimental): 33 subjects aged 65 years old with predisposition to cardiometabolic syndrome will consume 400ml of yogurt rich in cysteine, leucine and arginine (VP, vegetable proteins) only once during the visit
  Interventions: Behavioral: Vegetable proteins (VP) rich in leucine, cystein, arginine; Behavioral: Animal proteins (AP); Behavioral: No protein (T)
- Group/Cohort2 (Experimental): 33 subjects aged 65 years old with predisposition to cardiometabolic syndrome will consume 400ml of yogurt rich in animal proteins (AP) only once during the visit
  Interventions: Behavioral: Vegetable proteins (VP) rich in leucine, cystein, arginine; Behavioral: Animal proteins (AP); Behavioral: No protein (T)
- Group/Cohort3 (Placebo Comparator): 33 subjects aged 65 years old with predisposition to cardiometabolic syndrome will consume 400ml of yogurt without any proteins (T) only once during the visit
  Interventions: Behavioral: Vegetable proteins (VP) rich in leucine, cystein, arginine; Behavioral: Animal proteins (AP); Behavioral: No protein (T)

INTERVENTIONS:
Behavioral: Vegetable proteins (VP) rich in leucine, cystein, arginine — 33 volunteers will consume 400 ml of yogurt with vegetable proteins (VP) rich in leucine, cystein and arginine only once during the visit. At the beginning and the end of the intervention, exploration will be conducted at fasted state and at post-prandial state after the administration of vegetable proteins.
Behavioral: Animal proteins (AP) — 33 volunteers will consume 400 ml of yogurt with animal proteins (AP) rich in leucine, cystein and arginine only once during the visit. At the beginning and the end of the intervention, exploration will be conducted at fasted state and at post-prandial state after the administration of animal proteins.
Behavioral: No protein (T) — 33 volunteers will consume 400 ml of yogurt without any protein (T) rich in leucine, cystein and arginine only once during the visit. At the beginning and the end of the intervention, exploration will be conducted at fasted state and at post-prandial state after the administration of animal proteins.

SUMMARY:
By 2050, the expanding world population will consume two-thirds more animal protein than it consumes today. The increase in chronic diseases associated with the generalization of these consumption patterns tend to understand the place of meat in our diets. All these elements participate to the reduction of animal proteins in favor of vegetable proteins in our food. The elderly are particularly affected by malnutrition, the prevalence of protein-energy malnutrition increasing with age and promoting the onset of morbidities. Without care, it leads to the worsening of physiological phenomena linked to aging such as loss of muscle functionality (sarcopenia) or reduction in bone density (osteoporosis) and increases the risk of falls - the main cause of dependence. However, in France, protein consumption declines significantly with age, even though requirements appear to be greater for the elderly. It is therefore a major challenge for our societies to ensure that the aging of the population and the increase in life expectancy are not synonymous with a reduction in the physical and mental capacities of individuals. Thus, it is essential to ensure that the recommendations for reducing the intake of animal proteins in favor of vegetable proteins can be applied without risk to aging populations, in particular on the human body cardiovascular risk of these populations.

DETAILED DESCRIPTION:
This human dietary intervention study is a double blind, randomized, placebo controlled, cross over trial with 3 arms, carried out on subjects with predisposition to cardiometabolic syndrome (based on weight circumference, blood triglyceride or blood cholesterol, glycemia and hypertension). This study aims to demonstrate transient improvement in vascular endothelial function (with Flow Mediated Dilatation (FMD) as main criteria) with consumption of vegetable proteins (rich in leucine, cysteine and arginine) by comparison with animal proteins and with a control without proteins.

The 33 recruited participants will receive the 3 yogurts in a random order. For each subject, the study is divided into 4 visits.

To summarize: Visit 1 (D-7) = inclusion, Visit 2 (D0: treatment period N°1), Visit 3 (D28 : treatment period N°2), Visit 4 (D56 : treatment period N°3). The wash-out periods between treatment period (duration: 4 weeks) may be extended until 5 weeks for the convenience of participants.

The protocol includes a total of 4 visits to PIC/CIC Inserm 1405 of the Clermont-Fd University Hospital.

ELIGIBILITY:
Inclusion Criteria:

* Man or woman
* 65 years old and older (inclusive)
* At least 2 of the following 4 cardiometabolic factors:

  * Waist circumference ≥88 cm for women, and ≥94 cm for men
  * Fasting triglyceridemia >1,5 g/L OR HDL level < 40 mg/dl for men, and < 50 mg/dl for women
  * Fasting blood glucose ≥ 100 mg/dl
  * Systolic blood pressure >130mmHg ou diastolic > 85 mm Hg
* Accept not to change his lifestyle throughout the study
* Accept to consume the same meal the day before exploration days, making sure to exclude non-recommended foods and agreeing to detail its content in a food diary
* Ability to give informed consent to participate in research
* Affiliation to Social Security

Exclusion Criteria:

* Acute pathology (unstable or terminal pathology)
* Renal failure (clearance <40 mL / min)
* Asthma or chronic respiratory disease
* Systolic or diastolic blood pressure in the judgement of the investigator
* Diabetic (treated or not)
* Treated with chemotherapy
* Gastrointestinal, thyroid, cardiac or vascular illness in the judgement of the investigator
* Biological examination no compatible with the study in the judgement of the investigator
* Medical and/or surgical history no compatible with the study in the judgement of the investigator (previous cardiovascular events)
* AgHbS, AcHbc, HCV and HIV positive serology
* Concomitant treatment no compatible with the study in the judgement of the investigator
* Diet or change in body mass > 2 kg in the 30 days before the study
* Following a diet incompatible with the nutritional protocol (food intolerances, vegans, exclusion of certain food ingredients)
* Allergies to any of the components of the test meals
* Alcohol consumption> 2 glasses / day
* Current smokers (> 6 cigarettes per week)
* Subjects involved in another clinical trial or being in the exclusion period of another study or having received a total compensation greater than 4,500 euros over the 12 months preceding the start of the trial
* Subject benefiting from a legal protection measure (curatorship, guardianship, safeguard of justice)
* Refusal to participate

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 33 (Actual)
Dates: Start 2021-11-09 (Actual); Primary Completion 2022-06-07 (Actual); Study Completion 2022-06-07 (Actual)

PRIMARY OUTCOMES:
Brachial artery Flow Mediated Dilation (FMD) | Day 0 (V1) at T-30min
  The endothelial function will be assessed using the non-invasive ultrasound technique of flow mediated dilatation of the brachial artery. FMD measure is the percentage of dilation of brachial artery in response to a reactive hyperaemia induced by the release of a transient occlusion of the brachial artery realized.
Brachial artery Flow Mediated Dilation (FMD) | Day 0 (V1) at T180min
  The endothelial function will be assessed using the non-invasive ultrasound technique of flow mediated dilatation of the brachial artery. FMD measure is the percentage of dilation of brachial artery in response to a reactive hyperaemia induced by the release of a transient occlusion of the brachial artery realized between T-30min to T300min.
Brachial artery Flow Mediated Dilation (FMD) | Day 0 (V1) at T300min
  The endothelial function will be assessed using the non-invasive ultrasound technique of flow mediated dilatation of the brachial artery. FMD measure is the percentage of dilation of brachial artery in response to a reactive hyperaemia induced by the release of a transient occlusion of the brachial artery realized between T-30min to T300min.
Brachial artery Flow Mediated Dilation (FMD) | Day 28 (V2) at T-30min
  The endothelial function will be assessed using the non-invasive ultrasound technique of flow mediated dilatation of the brachial artery. FMD measure is the percentage of dilation of brachial artery in response to a reactive hyperaemia induced by the release of a transient occlusion of the brachial artery realized between T-30min to T300min.
Brachial artery Flow Mediated Dilation (FMD) | Day 28 (V2) at T180min
  The endothelial function will be assessed using the non-invasive ultrasound technique of flow mediated dilatation of the brachial artery. FMD measure is the percentage of dilation of brachial artery in response to a reactive hyperaemia induced by the release of a transient occlusion of the brachial artery realized between T-30min to T300min.
Brachial artery Flow Mediated Dilation (FMD) | Day 28 (V2) at T300min
  The endothelial function will be assessed using the non-invasive ultrasound technique of flow mediated dilatation of the brachial artery. FMD measure is the percentage of dilation of brachial artery in response to a reactive hyperaemia induced by the release of a transient occlusion of the brachial artery realized between T-30min to T300min.
Brachial artery Flow Mediated Dilation (FMD) | Day 56 (V3) at T-30min
  The endothelial function will be assessed using the non-invasive ultrasound technique of flow mediated dilatation of the brachial artery. FMD measure is the percentage of dilation of brachial artery in response to a reactive hyperaemia induced by the release of a transient occlusion of the brachial artery realized between T-30min to T300min.
Brachial artery Flow Mediated Dilation (FMD) | Day 56 (V3) at T180min
  The endothelial function will be assessed using the non-invasive ultrasound technique of flow mediated dilatation of the brachial artery. FMD measure is the percentage of dilation of brachial artery in response to a reactive hyperaemia induced by the release of a transient occlusion of the brachial artery realized between T-30min to T300min.
Brachial artery Flow Mediated Dilation (FMD) | Day 56 (V3) at T300min
  The endothelial function will be assessed using the non-invasive ultrasound technique of flow mediated dilatation of the brachial artery. FMD measure is the percentage of dilation of brachial artery in response to a reactive hyperaemia induced by the release of a transient occlusion of the brachial artery realized between T-30min to T300min.

SECONDARY OUTCOMES:
Rest flow by Flowmetry Laser Doppler (FLD) | Day 0 (V1), Day 28 (V2), Day 56 (V3)
  Vascular endothelial function in the micro-vascular compartment will be assessed using the measurement of the rest flow using laser-Doppler system at the level of the skin of the hand realized between T-30min to T300min.
Occlusion area by FLD | Day 0 (V1), Day 28 (V2), Day 56 (V3)
  Vascular endothelial function in the micro-vascular compartment will be assessed using the measurement of the occlusion area using laser-Doppler system at the level of the skin of the hand by following the response to a reactive hyperaemia induced by the release of a transient occlusion of the brachial artery (same stimulus as for FMD measurement) realized between T-30min to T300min.
Hyperaemia area by FLD | Day 0 (V1), Day 28 (V2), Day 56 (V3)
  Vascular endothelial function in the micro-vascular compartment will be assessed using the measurement of the hyperaemia area using laser-Doppler system at the level of the skin of the hand by following the response to a reactive hyperaemia induced by the release of a transient occlusion of the brachial artery (same stimulus as for FMD measurement) realized between T-30min to T300min.
Hyperaemia area / occlusion area ratio by FLD | Day 0 (V1), Day 28 (V2), Day 56 (V3)
  Vascular endothelial function in the micro-vascular compartment will be assessed using the ratio hyperaemia area / occlusion area determined by FLD realized between T-30min to T300min.
Maximal flow by FLD | Day 0 (V1), Day 28 (V2), Day 56 (V3)
  Vascular endothelial function in the micro-vascular compartment will be assessed using the measurement of the maximal flow using laser-Doppler system at the level of the skin of the hand by following the response to a reactive hyperaemia induced by the release of a transient occlusion of the brachial artery (same stimulus as for FMD measurement) realized between T-30min to T300min.
Hyperaemia half time by FLD | Day 0 (V1), Day 28 (V2), Day 56 (V3)
  Vascular endothelial function in the micro-vascular compartment will be assessed using the measurement of the hyperaemia half time using laser-Doppler system at the level of the skin of the hand by following the response to a reactive hyperaemia induced by the release of a transient occlusion of the brachial artery (same stimulus as for FMD measurement) realized between T-30min to T300min.
Reactive Hyperemia - Peripheral Arterial Tonometry (RH-PAT) | Day 0 (V1), Day 28 (V2), Day 56 (V3)
  Reactive hyperemia index (RHI) assessed by reactive hyperemia-peripheral arterial tonometry (RH-PAT) expressed as a percentage measures pulsatile fluctuations in digital volume in response to a reactive hyperaemia induced by the release of a transient occlusion realized between T-30min to T300min.
Plasma nitrite dosage | Day 0 (V1), Day 28 (V2), Day 56 (V3)
  Determination of nitrite plasma concentration (µmol/L) (a biomarker of endothelial activation) between T-90min to T360min.
Urine nitrite dosage | Day 0 (V1), Day 28 (V2), Day 56 (V3)
  Determination of nitrite urine concentration (µmol/L) (a biomarker of endothelial activation) between T-60min to T250min.
Plasma nitrate dosage | Day 0 (V1), Day 28 (V2), Day 56 (V3)
  Determination of nitrate plasma concentration (µmol/L) (a biomarker of endothelial activation) between T-90min to T360min.
Urine nitrate dosage | Day 0 (V1), Day 28 (V2), Day 56 (V3)
  Determination of nitrate urine concentration (µmol/L) (a biomarker of endothelial activation) between T-60min to T250min.
Plasma creatinine dosage | Day 0 (V1), Day 28 (V2), Day 56 (V3)
  Determination of creatinine plasma concentration (µmol/L) (a biomarker of chronic kidney disease) between T-90min to T360min.
Urine creatinine dosage | Day 0 (V1), Day 28 (V2), Day 56 (V3)
  Determination of creatinine urine concentration (µmol/L) (a biomarker of chronic kidney disease) between T-60min to T250min.
Plasma malondialdehyde (MDA) dosage | Day 0 (V1), Day 28 (V2), Day 56 (V3)
  Determination of MDA plasma concentration (nmol/L) (a biomarker of oxidative stress) between T-90min to T360min.
Urine malondialdehyde (MDA) dosage | Day 0 (V1), Day 28 (V2), Day 56 (V3)
  Determination of MDA urine concentration (nmol/L) (a biomarker of oxidative stress) between T-60min to T250min.
Plasma asymmetric dimethylarginine (ADMA) dosage | Day 0 (V1), Day 28 (V2), Day 56 (V3)
  Determination of ADMA plasma concentration (µmol/L) (a biomarker of cardiovascular disease) between T-90min to T360min.
Urine asymmetric dimethylarginine (ADMA) dosage | Day 0 (V1), Day 28 (V2), Day 56 (V3)
  Determination of ADMA urine concentration (µmol/L) (a biomarker of cardiovascular disease) between T-60min to T250min.
Plasma symmetric dimethylarginine (SDMA) dosage | Day 0 (V1), Day 28 (V2), Day 56 (V3)
  Determination of SDMA plasma concentration (µmol/L) (a biomarker of cardiovascular disease) between T-90min to T360min.
Urine symmetric dimethylarginine (SDMA) dosage | Day 0 (V1), Day 28 (V2), Day 56 (V3)
  Determination of SDMA urine concentration (µmol/L) (a biomarker of cardiovascular disease) between T-60min to T250min.
Plasma acetyl-lysine dosage | Day 0 (V1), Day 28 (V2), Day 56 (V3)
  Determination of acetyl-lysine plasma concentration (µmol/L) (a biomarker of vascular oxidative stress) between T-90min to T360min.
Urine symmetric acetyl-lysine dosage | Day 0 (V1), Day 28 (V2), Day 56 (V3).
  Determination of acetyl-lysine urine concentration (µmol/L) (a biomarker of vascular oxidative stress) between T-60min to T250min
Plasma N-epsilon-carboxy-methyl lysine (CML) dosage | Day 0 (V1), Day 28 (V2), Day 56 (V3).
  Determination of CML plasma concentration (pg/mL) (a biomarker of oxidative stress) between T-90min to T360min.
Urine N-epsilon-carboxy-methyl lysine (CML) dosage | Day 0 (V1), Day 28 (V2), Day 56 (V3).
  Determination of CML urine concentration (pg/mL) (a biomarker of oxidative stress) between T-60min to T250min.
Plasma N-epsilon-carboxy-ethyl lysine (CEL) dosage | Day 0 (V1), Day 28 (V2), Day 56 (V3).
  Determination of CEL plasma concentration (pg/mL) (a biomarker of oxidative stress) between T-90min to T360min.
Urine N-epsilon-carboxy-ethyl lysine (CEL) dosage | Day 0 (V1), Day 28 (V2), Day 56 (V3).
  Determination of CEL urine concentration (pg/mL) (a biomarker of oxidative stress) between T-60min to T250min.
Plasma alanine dosage | Day 0 (V1), Day 28 (V2), Day 56 (V3).
  Determination of alanine plasma concentration (µmol/L) between T-90min to T360min.
Urine alanine dosage | Day 0 (V1), Day 28 (V2), Day 56 (V3).
  Determination of alanine urine concentration (µmol/L) between T-60min to T250min.
Plasma arginine dosage | Day 0 (V1), Day 28 (V2), Day 56 (V3).
  Determination of arginine plasma concentration (µmol/L) between T-90min to T360min
Urine arginine dosage | Day 0 (V1), Day 28 (V2), Day 56 (V3).
  Determination of arginine urine concentration (µmol/L) between T-60min to T250min.
Plasma asparagine dosage | Day 0 (V1), Day 28 (V2), Day 56 (V3).
  Determination of asparagine plasma concentration (µmol/L) between T-90min to T360min
Urine asparagine dosage | Day 0 (V1), Day 28 (V2), Day 56 (V3).
  Determination of asparagine urine concentration (µmol/L) between T-60min to T250min.
Plasma aspartic acid dosage | Day 0 (V1), Day 28 (V2), Day 56 (V3).
  Determination of aspartic acid plasma concentration (µmol/L) between T-90min to T360min.
Urine aspartic acid dosage | Day 0 (V1), Day 28 (V2), Day 56 (V3).
  Determination of aspartic acid urine concentration (µmol/L) between T-60min to T250min.
Plasma cysteine dosage | Day 0 (V1), Day 28 (V2), Day 56 (V3).
  Determination of cysteine plasma concentration (µmol/L) between T-90min to T360min.
Urine cysteine dosage | Day 0 (V1), Day 28 (V2), Day 56 (V3).
  Determination of cysteine urine concentration (µmol/L) between T-60min to T250min
Plasma glutamic acid dosage | Day 0 (V1), Day 28 (V2), Day 56 (V3).
  Determination of glutamic acid plasma concentration (µmol/L) between T-90min to T360min.
Urine glutamic acid dosage | Day 0 (V1), Day 28 (V2), Day 56 (V3).
  Determination of glutamic acid urine concentration (µmol/L) between T-60min to T250min.
Plasma glutamine dosage | Day 0 (V1), Day 28 (V2), Day 56 (V3).
  Determination of glutamine plasma concentration (µmol/L) between T-90min to T360min
Urine glutamine dosage | Day 0 (V1), Day 28 (V2), Day 56 (V3).
  Determination of glutamine urine concentration (µmol/L) between T-60min to T250min.
Plasma glycine dosage | Day 0 (V1), Day 28 (V2), Day 56 (V3).
  Determination of glycine plasma concentration (µmol/L) between T-90min to T360min
Urine glycine dosage | Day 0 (V1), Day 28 (V2), Day 56 (V3).
  Determination of glycine urine concentration (µmol/L) between T-60min to T250min
Plasma histidine dosage | Day 0 (V1), Day 28 (V2), Day 56 (V3).
  Determination of histidine plasma concentration (µmol/L) between T-90min to T360min
Urine histidine dosage | Day 0 (V1), Day 28 (V2), Day 56 (V3).
  Determination of histidine urine concentration (µmol/L) between T-60min to T250min
Plasma isoleucine dosage | Day 0 (V1), Day 28 (V2), Day 56 (V3).
  Determination of isoleucine plasma concentration (µmol/L) between T-90min to T360min.
Urine isoleucine dosage | Day 0 (V1), Day 28 (V2), Day 56 (V3).
  Determination of isoleucine urine concentration (µmol/L) between T-60min to T250min.
Plasma leucine dosage | Day 0 (V1), Day 28 (V2), Day 56 (V3).
  Determination of leucine plasma concentration (µmol/L) between T-90min to T360min.
Urine leucine dosage | Day 0 (V1), Day 28 (V2), Day 56 (V3).
  Determination of leucine urine concentration (µmol/L) between T-60min to T250min.
Plasma lysine dosage | Day 0 (V1), Day 28 (V2), Day 56 (V3).
  Determination of lysine plasma concentration (µmol/L) between T-90min to T360min.
Urine lysine dosage | Day 0 (V1), Day 28 (V2), Day 56 (V3).
  Determination of lysine urine concentration (µmol/L) between T-60min to T250min.
Plasma methionine dosage | Day 0 (V1), Day 28 (V2), Day 56 (V3).
  Determination of methionine plasma concentration (µmol/L) between T-90min to T360min.
Urine methionine dosage | Day 0 (V1), Day 28 (V2), Day 56 (V3).
  Determination of methionine urine concentration (µmol/L) between T-60min to T250min.
Plasma phenylalanine dosage | Day 0 (V1), Day 28 (V2), Day 56 (V3).
  Determination of phenylalanine plasma concentration (µmol/L) between T-90min to T360min.
Urine phenylalanine dosage | Day 0 (V1), Day 28 (V2), Day 56 (V3).
  Determination of phenylalanine urine concentration (µmol/L) between T-60min to T250min.
Plasma proline dosage | Day 0 (V1), Day 28 (V2), Day 56 (V3).
  Determination of proline plasma concentration (µmol/L) between T-90min to T360min.
Urine proline dosage | Day 0 (V1), Day 28 (V2), Day 56 (V3).
  Determination of proline urine concentration (µmol/L) between T-60min to T250min.
Plasma serine dosage | Day 0 (V1), Day 28 (V2), Day 56 (V3).
  Determination of serine plasma concentration (µmol/L) between T-90min to T360min.
Urine serine dosage | Day 0 (V1), Day 28 (V2), Day 56 (V3).
  Determination of serine urine concentration (µmol/L) between T-60min to T250min.
Plasma threonine dosage | Day 0 (V1), Day 28 (V2), Day 56 (V3).
  Determination of threonine plasma concentration (µmol/L) between T-90min to T360min.
Urine threonine dosage | Day 0 (V1), Day 28 (V2), Day 56 (V3).
  Determination of threonine urine concentration (µmol/L) between T-60min to T250min.
Plasma tryptophan dosage | Day 0 (V1), Day 28 (V2), Day 56 (V3).
  Determination of tryptophan plasma concentration (µmol/L) between T-90min to T360min.
Urine tryptophan dosage | Day 0 (V1), Day 28 (V2), Day 56 (V3).
  Determination of tryptophan urine concentration (µmol/L) between T-60min to T250min.
Plasma tyrosine dosage | Day 0 (V1), Day 28 (V2), Day 56 (V3).
  Determination of tyrosine plasma concentration (µmol/L) between T-90min to T360min.
Urine tyrosine dosage | Day 0 (V1), Day 28 (V2), Day 56 (V3).
  Determination of tyrosine urine concentration (µmol/L) between T-60min to T250min.
Plasma valine dosage | Day 0 (V1), Day 28 (V2), Day 56 (V3).
  Determination of tyrosine plasma concentration (µmol/L) between T-90min to T360min.
Urine valine dosage | Day 0 (V1), Day 28 (V2), Day 56 (V3).
  Determination of tyrosine urine concentration (µmol/L) between T-60min to T250min.
Plasma Interleukin 6 (IL-6) dosage | Day 0 (V1), Day 28 (V2), Day 56 (V3).
  Determination of IL-6 plasma concentration (pg/ml) (a biomarker of inflammation and oxidative stress) between T-90min to T360min
Plasma Interleukin 1 bêta (IL-1β) dosage | Day 0 (V1), Day 28 (V2), Day 56 (V3).
  Determination of IL-1β plasma concentration (pg/ml) (a biomarker of inflammation and oxidative stress) between T-90min to T360min.
Plasma Monocyte Chemoattractant Protein-1 (MCP-1) dosage | Day 0 (V1), Day 28 (V2), Day 56 (V3).
  Determination of MCP-1 plasma concentration (pg/ml) (a biomarker of inflammation and oxidative stress) between T-90min to T360min.
Plasma Tumor Necrosis Factor alpha (TNFα) dosage | Day 0 (V1), Day 28 (V2), Day 56 (V3).
  Determination of TNFα plasma concentration (pg/ml) (a biomarker of inflammation and oxidative stress) between T-90min to T360min.
Plasma InterCellular Adhesion Molecule 1 (ICAM-1) dosage | Day 0 (V1), Day 28 (V2), Day 56 (V3).
  Determination of ICAM-1 plasma concentration (ng/ml) (a biomarker of endothelial activation) between T-90min to T360min.
Plasma E-Selectine dosage | Day 0 (V1), Day 28 (V2), Day 56 (V3).
  Determination of E-Selectine plasma concentration (ng/ml) (a biomarker of endothelial activation) between T-90min to T360min.
Transcriptome Sequencing of Peripheral Blood Mononuclear Cells | Day 0 (V1), Day 28 (V2), Day 56 (V3).
  Transcriptomic Analysis to quantify sets of genes involved in endothelial activation, oxidative stress, inflammation and cytokine expression between T-90 min to T360min.
Metabolome Sequencing of Plasma | Day 0 (V1), Day 28 (V2), Day 56 (V3).
  Untargeted Metabolomics to identify and quantify molecules involved in endothelial activation, oxidative stress, inflammation and cytokine expression between T-90 min to T360min.
Plasma Glucose dosage | Day 0 (V1), Day 28 (V2), Day 56 (V3).
  Determination of glucose plasma concentration (mg/dl) between T-90min to T360min.
Plasma triglycerides dosage | Day 0 (V1), Day 28 (V2), Day 56 (V3).
  Determination of triglycerides plasma concentration (mg/dl) between T-90min to T360min.
Plasma insulin dosage | Day 0 (V1), Day 28 (V2), Day 56 (V3).
  Determination of insulin plasma concentration (pmol/L) between T-90min to T360min
blood Peripheral Blood Mononuclear Cells (PBMC) count | Day 0 (V1), Day 28 (V2), Day 56 (V3).
  Determination of PBMC count (/mm3) and phenotyping between T-90min to T360min.
PBMC production of Reactive Oxygen Species (ROS) | Day 0 (V1), Day 28 (V2), Day 56 (V3).
  Assessment of the ROS level (between T-90min to T360min) produced by isolated PBMC following oxidative stress induction.
Questionnaire of acceptability | Day 0 (V1), Day 28 (V2), Day 56 (V3).
  Acceptability was assessed by a 9-point time scale where "1" means a very poor acceptability and "9" means a very good acceptability.

CONTACTS AND LOCATIONS:
Overall Officials: Gisèle PICKERING, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU clermont-ferrand, Clermont-Ferrand, France

REFERENCES:
- [Derived] Dimina LJ, Leray V, Voute M, David J, Blavignac C, Farges MC, Rossary A, Tsikas D, Remond D, Pickering G, Mariotti F. Dietary Protein in a Challenge Meal Does Not Alleviate Postprandial Impairments in Vascular Endothelial Function in Healthy Older Adults with Cardiometabolic Risk: A Randomized Crossover-Controlled Trial. J Nutr. 2024 Dec;154(12):3664-3680. doi: 10.1016/j.tjnut.2024.10.018. Epub 2024 Oct 16. PMID 39424070